CLINICAL TRIAL: NCT04882228
Title: A Multicenter, Double-blind, Randomized, Active Controlled, Parallel Group, Non-inferiority Phase 4 Study to Evaluate Efficacy and Safety of Entelon Tab.150mg in Patients With Chronic Venous Disease(CVD)
Brief Title: Phase 4 Study to Evaluate Efficacy and Safety of Entelon Tab.150mg in Patients With Chronic Venous Disease(CVD)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hanlim Pharm. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HL_ENTL_401
Record Dates: First submitted 2021-05-06; First posted 2021-05-11 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-04

CONDITIONS: Chronic Venous Disease
MeSH Terms: interventions — S 5682

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Entelon Tab.150mg (Experimental)
  Interventions: Drug: Entelon Tab.150mg; Drug: Placebo of Venitol Tab.
- Venitol tab. (Active Comparator)
  Interventions: Drug: Venitol Tab.; Drug: Placebo of Entelon Tab.150mg

INTERVENTIONS:
Drug: Entelon Tab.150mg — twice daily for 8 weeks
  Other Names: Vitis Vinifera Seed Dreid Extract 150mg
  Arms: Entelon Tab.150mg
Drug: Venitol Tab. — twice daily for 8 weeks
  Other Names: Purified and Micronized Flavonoid Fraction 500mg
  Arms: Venitol tab.
Drug: Placebo of Venitol Tab. — twice daily for 8 weeks (with Entelon Tab.150mg. It is for the masking.)
  Arms: Entelon Tab.150mg
Drug: Placebo of Entelon Tab.150mg — twice daily for 8 weeks(with Venitol Tab. It is for the masking.)
  Arms: Venitol tab.

SUMMARY:
This clinical trial is a multi-center, double-blind, randomized, active controlled , parallel design, non-inferiority phase 4 study to evaluate the efficacy and safety of Entelon 150mg in 278 patients with chronic venous disease.

DETAILED DESCRIPTION:
This study is to prove that Entelon tab. 150mg is non-inferior in clinical efficacy and safety compared to Venitol tab. for 8 weeks in patients suffering from chronic venous disease.

ELIGIBILITY:
Inclusion Criteria:

1. 19 years ≤ age ≤ 80 years
2. Those who are diagnosed as CEAP Classification Class 1 ~ Class 3
3. Those who have the Venous Duplex ultrasonography result at least one of the following

   * reflux more than 1 second in Femoral vein or Popliteal vein
   * reflux more that 0.5 second in GSV or SSV or Accessory saphenous vein or perforating vein or calf vein
4. Those who have completed the washout period as following until the baseline, including the screening period

   * Analgesic, corticosteroids, anti-inflammatory drugs: at least 2 weeks
5. Those who provide written consent voluntarily to participate in this clinical trial

Exclusion Criteria:

1. Those who must wear compression stockings
2. Those who have obstruction of the peripheral arteries of the lower extremities
3. Those who have asymptomatic varicose veins
4. Those who have acute deep vein thrombosis
5. Those who have frequent lower extremity pain due to neuropathy
6. Varicose vein surgery patient or prospective person (if surgery was done more than 1 year prior to the time of screening, recruitment is possible)
7. Those who have systemic disease that causes edema or thrombosis
8. Those who have a history of malignant tumors within 5 years prior to the time of screening
9. Those who have severe renal dysfunction at the time of screening (serum creatinine ≥ 2 x upper limit of normal)
10. Those who have severe liver dysfunction at the time of screening (AST or ALT ≥ 3 x upper limit of normal)
11. Those who are required to receive diuretics, analgesics, corticosteroids, anti-inflammatory drugs, or contraindications that may affect the outcome of this clinical trial during the clinical trial period
12. Those who have a history of significant mental illness, alcohol abuse
13. Patients who have an allergy to investigational product or any of its excipients
14. Patients who participated in other clinical trials within 12 weeks prior to the date of screening
15. Pregnant or lactating woman
16. Those who do not agree to use an effective method of contraception
17. Individual considered by the investigator to be ineligible for study participation

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 278 (Estimated)
Dates: Start 2021-01-28 (Actual); Primary Completion 2022-02-28 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
CIVIQ-20 questionnaire score change | 8week(Visit 4)
  Change at week 8 of treatment with the drug from baseline(day 0) in CIVIQ-20 questionnaire score

SECONDARY OUTCOMES:
CIVIQ-20 questionnaire score change | 4week(Visit 3)
  Change at week 4 of treatment with the drug from baseline(day 0) in CIVIQ-20 questionnaire score
AVVQ questionnaire score change | 4week(Visit 3), 8week(Visit 4)
  Change at week 4, 8 of treatment with the drug from baseline(day 0) in AVVQ questionnaire score
100mm VAS score change of leg heaviness, leg pain, leg cramps | 4week(Visit 3), 8week(Visit 4)
  Change at week 4, 8 of treatment with the drug from baseline(day 0) in symptoms of leg heaviness, leg pain, leg cramps thorugh 100mm VAS score
Venous clinical severity score change | 4week(Visit 3), 8week(Visit 4)
  change at week 4, 8 of treatment with the drug from baseline(day 0) in Venous clinical severity score
change in the circumference of the leg due to edema | 8week(Visit 4)
  change at week 8 of treatment with the drug from baseline(day 0) in leg circumference

CONTACTS AND LOCATIONS:
Locations (1):
- Bundang Seoul University Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No